CLINICAL TRIAL: NCT01263587
Title: Observational Study of Persons With Hepatitis B Virus Infection in North America (Cohort Study)
Brief Title: Hepatitis B Research Network Adult Cohort Study
Acronym: HBRN
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Anna Lok, Study Chair, University of Michigan
Other Study IDs: DK082864; U01DK082864 (NIH); U01DK082843 (NIH); U01DK082866 (NIH); U01DK082863 (NIH); U01DK082867 (NIH); U01DK082871 (NIH); U01DK082872 (NIH); U01DK082874 (NIH); U01DK082919 (NIH); U01DK082923 (NIH); U01DK082927 (NIH); U01DK082943 (NIH); U01DK082944 (NIH); P30DK050306 (NIH); A-DK-3002-001 (Other Grant/Funding Number: Interagency agreement); M01RR000040 (NIH); UL1TR000058 (NIH); UL1TR000004 (NIH); UL1RR024986 (NIH); UL1TR001111 (NIH); NCT01306071 (obsolete NCT alias)
Record Dates: First submitted 2010-12-14; First posted 2010-12-20 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HBV; Cohort Study
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy tissue, blood (serum, plasma, and DNA)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to describe participants with hepatitis B virus (HBV) infection and identify factors that may cause the disease to activate or worsen.

DETAILED DESCRIPTION:
Aims

* Primary Aim:

  o To describe participants with hepatitis B virus (HBV) infection in a prospective cohort in the United States (US) and Canada and identify predictors of disease activation and progression
* Secondary Aims:

  * To describe clinical, virological, and immunological characteristics of participants with HBV in the US and Canada
  * To evaluate changes in HBV infection status and quantitative hepatitis B surface antigen (HBsAg) levels and factors associated with those changes
  * To verify whether a baseline HBsAg below 1,000 IU/mL and HBV DNA below 1,000 IU/mL is an accurate predictor of people who are, or who will become, inactive carriers, defined as people who are HBsAg positive, hepatitis B "e" antigen (HBeAg) negative, have normal Alanine transaminase (ALT) and HBV DNA under 1,000 IU/mL on at least two occasions over a period of at least 6 months
  * To develop a bank of biospecimens (e.g., serum, plasma, DNA, lymphocytes, liver tissue) obtained from participants with HBV infection
  * To identify participants with HBV infection who are potential candidates in one of the treatment studies to be conducted by the Hepatitis B Research Network (HBRN)
  * To describe the natural history of hepatitis B infection in pregnancy including the frequency of, and clinical and virological characteristics associated with, hepatic flares during pregnancy and post-partum.

ELIGIBILITY:
The study population will be recruited from multi-site clinical centers in the United States and Canada including primary care hospitals and community centers.

Inclusion criteria

* Written informed consent
* At least 18 years of age
* Hepatitis B surface antigen (HBsAg) positive and either:

  * Pregnant
  * Anti-Hepatitis D positive
  * Diagnosed with acute Hepatitis B infection or experiencing a hepatitis flare
  * Immune tolerant or immune active phenotype
  * Potentially eligible for the Immune Regulation and Costimulation in Natural History of Chronic Hepatitis B ancillary study (NCT01298037).

Exclusion Criteria:

* Hepatic decompensation
* Hepatocellular carcinoma (HCC)
* Liver transplantation
* Current hepatitis B antiviral treatment (except pregnant women and patients who are anti-HDV positive)
* Known Human immunodeficiency virus (HIV) co-infection (patients with Hepatitis D (HDV) or Hepatitis C (HCV) co-infection are not excluded).
* Medical or social condition which in the opinion of the investigator will interfere with or prevent follow-up per protocol
* Unable or unwilling to return for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from multi-site clinical centers in the United States and Canada including primary care hospitals and community centers.
Sampling Method: Non-Probability Sample
Enrollment: 2051 (Actual)
Dates: Start 2010-12; Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Hepatitis Exacerbation marked by alanine aminotransferase (ALT) Flare | up to 288 weeks
  A flare is defined as serum ALT greater than or equal to 10 times the upper limit of normal which corresponds to 300 IU/L in males or 200 IU/L in females. This definition will also be applied to hepatitis B surface antigen (HBsAg) positive pregnant women whose ALT levels increase during pregnancy or postpartum. Once a flare is detected, participants will be followed more closely until its resolution.
Antigen loss: e and s | up to 288 weeks
  Loss of these viral markers may be associated with appearance of corresponding antibodies in serum (anti-HBe or anti-HBs). HBsAg loss appears to represent a "cure" of HBV infection and is associated with reduction, but not necessarily elimination, of the risk of future complications, such as Hepatocellular carcinoma (HCC) which may occur, particularly in those who lose HBsAg at an older age (after 50 years) or after the development of cirrhosis. When HBeAg or HBsAg loss occurs, participants will be followed more closely initially and then return to the regular follow-up schedule.
Cirrhosis | up to 288 weeks
  Once cirrhosis is diagnosed, follow-up will include hepatocellular carcinoma (HCC) surveillance. HCC surveillance will also be performed in non-cirrhotic participants who meet American Association for the Study of Liver Disease guidelines criteria.
Hepatic decompensation | up to 288 weeks
  Development of hepatic decompensation will be defined by any of the following events:
  * Ascites or hepatic hydrothorax
  * Variceal or portal hypertensive bleeding
  * Hepatic encephalopathy
  * Child-Turcotte-Pugh (CTP) score of 7 or above
  It is anticipated that there will be a small number of participants who will develop hepatic decompensation during follow-up.
Hepatocellular carcinoma (HCC) | up to 288 weeks
  Hepatocellular carcinoma (HCC) may be detected by routine surveillance or may become clinically apparent. The diagnosis of HCC will be made using the American Association for the Study of Liver Disease criteria.
Death | up to 288 weeks
  Death may occur related to liver disease (typically hepatic decompensation or Hepatocellular carcinoma) or may occur unrelated to hepatitis B or liver disease. Date and cause of death will be recorded.
Liver transplantation | up to 288 weeks
  Liver transplantation will be recorded upon notification. Date of transplantation, indication for transplantation, and occurrence of incidental Hepatocellular carcinoma (HCC) will be recorded. Follow-up ends with liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Belle, PhD, Principal Investigator — University of Pittsburgh
Locations (21):
- United States (20):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - The Queen's Medial Center, Honolulu, Hawaii
  - NIH Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
- Toronto Western Hospital Liver Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lisker-Melman M, King WC, Ghany MG, Chung RT, Hinerman AS, Cloherty GA, Khalili M, Jain MK, Sulkowski M, Sterling RK. Human immunodeficiency virus coinfection differentially impacts hepatitis B virus viral markers based on hepatitis Be antigen status in patients with suppressed viremia. J Viral Hepat. 2023 Aug;30(8):700-709. doi: 10.1111/jvh.13857. Epub 2023 Jun 6. PMID 37278302
- [Derived] Sterling RK, Wahed AS, Cloherty G, Hoofnagle JH, Lee WM; Hepatitis B Research Network Investigators. Acute Hepatitis B Virus Infection in North American Adults. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1881-1892.e4. doi: 10.1016/j.cgh.2022.09.004. Epub 2022 Sep 16. PMID 36116752
- [Derived] Khalili M, Kleiner DE, King WC, Sterling RK, Ghany MG, Chung RT, Bhan AK, Rosenthal P, Lisker-Melman M, Ramachandran R, Lok AS; ; and the Hepatitis B Research Network (HBRN). Hepatic Steatosis and Steatohepatitis in a Large North American Cohort of Adults With Chronic Hepatitis B. Am J Gastroenterol. 2021 Aug 1;116(8):1686-1697. doi: 10.14309/ajg.0000000000001257. PMID 33840726
- [Derived] Evon DM, Lin HS, Khalili M, Fontana RJ, Yim C, Wahed AS, Fried MW, Hoofnagle JH; Hepatitis B Research Network (HBRN). Patient-reported outcomes in a large North American cohort living with chronic hepatitis B virus: a cross-sectional analysis. Aliment Pharmacol Ther. 2020 Feb;51(4):457-468. doi: 10.1111/apt.15618. Epub 2020 Jan 14. PMID 31943262
- [Derived] Di Bisceglie AM, King WC, Lisker-Melman M, Khalili M, Belle SH, Feld JJ, Ghany MG, Janssen HLA, Lau D, Lee WM, Ling SC, Cooper S, Rosenthal P, Schwarz KB, Sterling RK, Teckman JH, Terrault N; Hepatitis B Research Network (HBRN). Age, race and viral genotype are associated with the prevalence of hepatitis B e antigen in children and adults with chronic hepatitis B. J Viral Hepat. 2019 Jul;26(7):856-865. doi: 10.1111/jvh.13104. Epub 2019 May 2. PMID 30974509
- [Derived] Khalili M, Shuhart MC, Lombardero M, Feld JJ, Kleiner DE, Chung RT, Terrault NA, Lisker-Melman M, Sanyal A, Lok AS; Hepatitis B Research Network (HBRN); Harvard Consortium. Relationship Between Metabolic Syndrome, Alanine Aminotransferase Levels, and Liver Disease Severity in a Multiethnic North American Cohort With Chronic Hepatitis B. Diabetes Care. 2018 Jun;41(6):1251-1259. doi: 10.2337/dc18-0040. Epub 2018 Mar 29. PMID 29599296
- [Derived] Di Bisceglie AM, Lombardero M, Teckman J, Roberts L, Janssen HL, Belle SH, Hoofnagle JH; Hepatitis B Research Network (HBRN). Determination of hepatitis B phenotype using biochemical and serological markers. J Viral Hepat. 2017 Apr;24(4):320-329. doi: 10.1111/jvh.12643. Epub 2016 Dec 5. PMID 27917600
- See also: The Hepatitis B Research Network study web site — http://www.hepbnet.org/